CLINICAL TRIAL: NCT00188266
Title: Prospective Phase I/II Study of Adjuvant Radiochemotherapy for Gastric Cancer
Brief Title: Study of Adjuvant Radiochemotherapy for Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 02-0134-C
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-Fluorouracil (5FU) and Cisplatin with Radiation (Experimental)
  Interventions: Drug: cisplatinum combined with infusional fluorouracil (5 FU)

INTERVENTIONS:
Drug: cisplatinum combined with infusional fluorouracil (5 FU) — Continuous 5FU via intravenous PICC line + 4 doses of Cisplatin every 2 weeks

SUMMARY:
In 1991, the South West Oncology Group (SWOG) conducted a randomized study of adjuvant chemotherapy (5-fluorouracil and folinic acid) with concurrent radiation (4500 cGy/25 fractions) versus surgery alone for patients with completely resected gastric carcinoma.

This landmark study showed the benefit of adjuvant treatment for gastric cancer and radically changed the treatment of this disease. However, the resulting standard treatment has severe acute toxicity, and despite this advance, 50% of patients still die of gastric cancer. The investigators hope to develop a modified protocol using active chemotherapy agents, but with reduced acute toxicity. Such an approach could ultimately be studied against the current SWOG approach to determine whether or not the addition of cisplatinum improves efficacy.

Patients who decide to participate in the study will receive a chemotherapy drug called 5-Fluorouracil (5FU)through an intravenous catheter continuously over 12 weeks. Patients will not be admitted to hospital to receive the chemotherapy but will need to wear a waist pack to carry a small pump that will deliver the medication. They will however need to make regular visits to have their medication bags changed. Patients will also receive Cisplatin intravenously every 2 weeks for 4 doses. In addition, patients will also receive radiation to their stomach, lymph nodes, and the area where they had their surgery. This study also comprise of a questionnaire for us to see how patient's cancer and treatment is affecting their quality of life. Patients will have regular follow-up by their physicians.

ELIGIBILITY:
Inclusion Criteria:

* R0 resection (no microscopic residual) of adenocarcinoma of stomach or gastroesophageal (GE) junction, prior to starting chemotherapy and radiation
* Tumor must not extend more than 2 cm along the esophagus; bulk of the tumor must be in the stomach.
* Adequate pre-operative cross-sectional imaging (computed tomography [CT] or magnetic resonance imaging [MRI])
* International Union Against Cancer (UICC)/American Joint Committee on Cancer (AJCC) Stage IB - IV, excluding patients with metastatic disease (T1N1, T2N0 to T4N1, N2, and any T, N3). T2N0 eligible only if disease extends beyond muscularis propria.
* No previous abdominal radiotherapy or contraindication to radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Adequate major organ function
* Nutritional intake of at least 1500 calories per day at nutrition assessment
* Treatment started within 20-90 days post-op of surgery date.
* Informed consent

Exclusion Criteria:

* Less than 70 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2002-08 (Actual); Primary Completion 2013-12-19 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Phase I and II: Acute toxicity: assessed according to National Cancer Institute of Canada (NCIC) and Radiation Therapy Oncology Group (RTOG) toxicity assessment criteria. | 10 years
Phase II: Comparison of acute toxicity rates with those observed in their previous study of 20 patients treated similarly to the SWOG INT 0116 protocol. | 10 year

SECONDARY OUTCOMES:
Monitor 1 and 2 year local recurrence | 10 years
Survival and disease-specific survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jolie Ringash, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada